CLINICAL TRIAL: NCT05932953
Title: Skin Tolerance of Medical Devices for Diabetes Monitoring and Treatment in Children With Type 1 Diabetes, an Observational, Retrospective, Single-center Study.
Brief Title: Skin Tolerance of Medical Devices for Diabetes Monitoring and Treatment in Children With Type 1 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, RENARD Emeline, principal investigator, Central Hospital, Nancy, France
Other Study IDs: 2022PI015
Record Dates: First submitted 2022-05-09; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Cutaneous Allergy; Diabetes Mellitus, Type 1; Atopic Disorders
Keywords: diabetes mellitus, type 1; cutaneous allergy; atopic disorders
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionary — questionary about cutaneous tolerance

SUMMARY:
In view of the emergence over the last few years of adverse skin reactions caused by diabetes monitoring and treatment devices, which have become essential to the optimal management of these patients, it is necessary to determine the real prevalence of these side effects.

Here the investigators performed a prospective study about prevalence of skin reactions in a group of children with type 1 diabetes.

DETAILED DESCRIPTION:
Justification :

* The incidence of type 1 diabetes in children is increasing every year.
* The use of blood glucose sensors has a positive impact on blood glucose control by limiting glucose variability, reducing hypoglycemia and improving long-term blood glucose control.
* The first cases of allergic contact dermatitis secondary linked to the use of an insulin pump were identified in 1995.
* Several recent studies report a high prevalence of allergic contact dermatitis caused to blood glucose sensors, but these studies are conducted on small samples and in most cases these samples include both adults and children.
* The actual prevalence of children with adverse skin reactions secondary to their diabetes monitoring and treatment devices is probably underestimated
* IBOA was the first responsible allergen identified in 2016. It is the most common allergen responsible for these allergic contact dermatitis3, but other allergens have also been identified recently.
* It is difficult to say how many diabetic patients have ever developed a contact allergy to IBOA, or other acrylates, in their skin devices. Typically, the reaction does not appear until after prolonged use, usually after several months.
* Very few studies have looked at the impact on children's quality of life. In view of the emergence over the last few years of adverse skin reactions caused by diabetes monitoring and treatment devices, which have become essential to the optimal management of these patients, it is necessary to determine the real prevalence of these side effects. The research of risk factors associated with the appearance of these lesions, as well as the impact on patient's quality of life is essential, so as to be able to prevent them and treat them if necessary.

General outline of the study:

Epidemiological, observational, cross-sectional, retrospective study carried out on a sample of the target population after collecting data both on questionnaires and in the patients' medical files. The questionnaires and the data sought in the patients' files will be collected over a period of 1 year, after obtaining the parents' non objection. The questionnaires will be distributed by the medical and paramedical team of the pediatric diabetes service of the Nancy CHRU. They will be hand-delivered to the physician leading the quarterly follow-up visit of the child's. No additional consultation will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

* -Children under 18 years of age
* Diabetic (type 1) for more than one month at the time of data collection and questionnaire completion
* Wearing an insulin pump and/or a blood glucose sensor.

Exclusion Criteria:

* - Parental refusal to participate in the study.
* Other types of diabetes than type 1 (type 2 diabetes, MODY...)
* Diabetes diagnosed less than one month before data collection and questionnaire completion

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children aged 0 to 18 years, type 1 diabetics, followed at the CHRU of Nancy and wearing a blood glucose sensor and/or an insulin pump.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of children,with current skin intolerance (eczema symptoms measured by questionnaire) to an insulin pump and/or blood glucose sensor assessed by an autoquestionnary. | 24 months
  Prevalence of of children, under 18 years of age, with type 1 diabetes with current skin intolerance to an insulin pump and/or blood glucose sensor. Pruritus, erythema, scaling, vesicles, and scratching lesions that appear at the infusion set site location of blood glucose sensors and insulin pumps are considered skin intolerance. (evaluated by questionnaire)

SECONDARY OUTCOMES:
- Prevalence of skin side effects (eczema symptoms measured by questionnaire) for sensors and insulin pumps each one taken. | 24 months
  - Prevalence of skin side effects (eczema symptoms measured by questionnaire) for sensors and insulin pumps each one taken.
Search for risk factors associated with skin side effect | 24 months
  Odds ratio calculated for risk factors suspected in skin reaction

CONTACTS AND LOCATIONS:
Overall Officials: Emeline RENARD, PhD, Principal Investigator — CHRU Nancy
Locations (1):
- CHRU Nancy, Nancy, France